CLINICAL TRIAL: NCT03238586
Title: HIV/AIDS & Alcohol-Related Outcomes: Translational Evidence-Based Interventions
Acronym: WELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Patricia Molina, Richard Ashman, PhD Professor and Head Department of Physiology; Director Alcohol and Drug Abuse Center of Excellence, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WELL; 1U01AA021995-01 (NIH)
Record Dates: First submitted 2017-07-31; First posted 2017-08-03 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: HIV/AIDS
Keywords: hiv; aids; alcohol; health; knowledge; motivation; skills; behavior
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Behavior

ARMS (2):
- WELL Program (Experimental): Five-week treatment program that aims to improve knowledge, motivation, and skills. It is designed to motivate participants to take their medications routinely, improve the quality of life for those living with HIV, and decrease risky behaviors that may lead to HIV transmission.
  Interventions: Behavioral: WELL Program
- Standard of Care (No Intervention): Five-week standard of care program.

INTERVENTIONS:
Behavioral: WELL Program
  Arms: WELL Program

SUMMARY:
A clinical study for patients with HIV that investigates the best way to reduce HIV transmission risk, and to improve the overall health of people living with HIV/AIDS. Participants will complete four assessments over the course of one year and will be randomly assigned to a five-week treatment program.

DETAILED DESCRIPTION:
The main purpose of this research study is to investigate the best way to reduce HIV transmission risk and to improve the overall health of people living with HIV/AIDS. This study tests an intervention program that aims to improve knowledge, motivation, and skills. The intervention program is designed to motivate participants to take their medications routinely, improve the quality of life for those living with HIV, and decrease risky behaviors that may lead to HIV transmission.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Recent alcohol use

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Viral load | Change from baseline at 3 months, 6 months and 1 year
  The primary outcome measure will be disease progression or more specifically, the proportion of patients achieving viral suppression.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Molina, MD, PhD, Principal Investigator — Louisiana State University Health Sciences Center
Locations (1):
- University Medical Center New Orleans Infectious Disease Services, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided